CLINICAL TRIAL: NCT04656691
Title: At-Home Infusion Using Bamlanivimab in Participants With Mild to Moderate COVID-19
Acronym: UNITED
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: In April 2021 FDA revoked the Emergency Use Authorization after determining that the known and potential benefits of bamlanivimab, when administered alone, no longer outweigh the known and potential risks for its authorized use.
Sponsor: Daniel Griffin (Industry)
Collaborators: Eli Lilly and Company (Industry); Optum, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Daniel Griffin, Daniel Griffin, MD PhD CTropMed CTH, UnitedHealth Group
Organization: UnitedHealth Group (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0081_
Record Dates: First submitted 2020-12-04; First posted 2020-12-07 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: COVID19; bamlanivimab; UnitedHealth
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab

STUDY DESIGN:
Intervention Model Description: Participants that test positive for COVID-19 may be eligible to receive an in-home infusion of bamlanivimab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with COVID-19 (Experimental): Participants testing positive for COVID-19 may be eligible to receive a one-time dose of bamlanivimab 700 mg, delivered via infusion through the vein, lasting around 60 minutes. This infusion will be done in-home and administered by a registered nurse.
  Interventions: Drug: bamlanivimab

INTERVENTIONS:
Drug: bamlanivimab — Participants that test positive for COVID-19 may be eligible to receive an in-home infusion of bamlanivimab by a registered nurse. This infusion will last approximately 1 hour followed by 1 hour of observation.

SUMMARY:
This is an open-label, pragmatic, single-dose study using matched controls in participants with mild to moderate COVID-19. Participants will track for developing symptoms while at home and upon reporting of symptoms will test for COVID-19. If positive for COVID-19, a one-time at-home infusion of Bamlanivimab (LY3819253) will be provided by Optum Infusion. Participants will then track for 28 days to assess for any additional medical care needed or if hospitalization was required.

ELIGIBILITY:
Inclusion Criteria:

* UnitedHealthcare member
* confirmed COVID-19 positive
* located in an area where Bamlanivimab (LY3819253) is available for infusion

Exclusion Criteria:

* current (from first symptom report) hospitalization for COVID-19
* prior administration of Bamlanivimab or other COVID-19 therapies
* previous COVID-19 diagnosis
* prior receipt of a COVID-19 vaccine
* not authorized for patient use per the EUA

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 139 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Griffin, MD, PHD, Principal Investigator — ProHealth New York - UnitedHealth Group
Locations (1):
- QueryLab, Minnetonka, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share participant level data with other projects or researchers.

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The treatment group was identified by the following inclusion and exclusion criteria once they report symptoms and test positive of COVID-19. They were offered an in-home infusion of 700 mg Bamlanivimab by a nurse within 10 days of their symptom onset if they consent. Email/mail invitations to consider participation will be sent to those who qualify to consider joining to track for symptoms (located in an area where Bamlanivimab (LY3819253) is currently available)
Pre-assignment Details: Inclusion:
  * Age 65+, confirmed SARS-CoV-2 positive, located in an area where Bamlanivimab (LY3819253) is available for infusion,
  * Have mild or moderate COVID-19 symptoms OR
  * Individuals who are at high risk for progression to severe COVID-19 in the Emergency Use Authorization (EUA) of Bamlanivimab (page 4 at the EUA; EUA revoked on April 16, 2021)
  Exclusion Criteria:
  * Current (from first symptom report) hospitalization for COVID-19
  * Prior administration of Bamlanivimab
Groups:
- Treatment: Participants With COVID-19: Participants testing positive for COVID-19 may be eligible to receive a one-time dose of bamlanivimab 700 mg, delivered via infusion through the vein, lasting around 60 minutes. This infusion will be done in-home and administered by a registered nurse followed by 1 hour of observation..
Period: Overall Study
Arm/Group | Treatment: Participants With COVID-19
Started | 139
Completed | 138
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With COVID-19
Number analyzed (Participants) | 139
Age, Customized [Count of Participants; unit: Participants] — Count percentage of participants aged 64 years and older in customized age groups Population: 139 infusions were started with 138 fusions being completed - that is the discrepancy between the number of infusions started (139) and the number completed (138) and the number considered evaluable (only completed infusions at 138)
  Participants
    64 years or younger | 4
    65 years to 69 years | 51
    70 years to 74 years | 46
    75 years to 79 years | 21
    80 years or older | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Pacific Islander | 0
  Black or African American | 3
  White | 72
  Other | 2
  Race Unknown or Not Reported | 62
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Ethnicity Unknown or Not Reported | 139
Days since COVID-19 symptom onset (count) [Count of Participants; unit: Participants] — This measure describes when study participants got an at-home infusion since COVID-19 symptom onset in days. Population: Date of COVID-19 symptom onset was confirmed for 128 participants of the total 139 participants
  Participants
    Equal to or less than 8 days since COVID-19 symptom onset | 128
    Greater than 8 days since COVID-19 symptom onset | 1
    Unknown | 10
Days since COVID-19 symptom onset (mean) [Mean (Standard Deviation); unit: Days] — Population: Date of COVID-19 symptom onset was not available for all participants
  Days
    number analyzed (Participants) | 129
    (all) | 3.7 (2.24)
Elixhauser comorbidity score (Mean) [Mean (Standard Deviation); unit: units on a scale] — It is a weighted score of the 29 Elixhauser comorbid conditions designed to predict risk of in-hospital mortality or 30-day, all-cause readmission (Moore et al., 2017). The conditions include deficiency anemia, depression, uncomplicated diabetes, diabetes with chronic complications, etc. We used the 2019 version for the outcome of 30-day, all-cause readmission by Agency for Healthcare Research and Quality (AHRQ). The Elixhauser score ranges from -4 to 219, with higher scores indicating a higher patient comorbidity Population: Medical Record and Claims data were not available for all infused participants to establish the Elixhauser comorbidity score. The score provides context for outcome measures and was not required to determine eligibility
  units on a scale
    number analyzed (Participants) | 82
    (all) | 9.3 (13.09)
Elixhauser conditions [Count of Participants; unit: Participants] — Population: Medical Record and Claims data were not available for all infused participants to identify Elixhauser conditions. The score provides context for outcome measures and was not required to determine eligibility. Some participants had multiple Elixhauser conditions
  Participants
    Acquired Immune Deficiency Syndrome: number analyzed (Participants) | 82
    Acquired Immune Deficiency Syndrome | 0
    Alcohol Abuse: number analyzed (Participants) | 82
    Alcohol Abuse | 2
    Deficiency Anemia: number analyzed (Participants) | 82
    Deficiency Anemia | 14
    Rheumatoid arthritis/collagen vascular diseases: number analyzed (Participants) | 82
    Rheumatoid arthritis/collagen vascular diseases | 1
    Chronic blood loss anemia: number analyzed (Participants) | 82
    Chronic blood loss anemia | 2
    Congestive heart failure: number analyzed (Participants) | 82
    Congestive heart failure | 5
    Chronic pulmonary disease: number analyzed (Participants) | 82
    Chronic pulmonary disease | 12
    Coagulopathy: number analyzed (Participants) | 82
    Coagulopathy | 4
    Depression: number analyzed (Participants) | 82
    Depression | 9
    Diabetes, Uncomplicated: number analyzed (Participants) | 82
    Diabetes, Uncomplicated | 17
    Diabetes, With Chronic Complications: number analyzed (Participants) | 82
    Diabetes, With Chronic Complications | 12
    Drug Abuse: number analyzed (Participants) | 82
    Drug Abuse | 1
    Hypertension, Complicated or Uncomplicated: number analyzed (Participants) | 82
    Hypertension, Complicated or Uncomplicated | 51
    Hypothyroidism: number analyzed (Participants) | 82
    Hypothyroidism | 13
    Liver Disease: number analyzed (Participants) | 82
    Liver Disease | 3
    Lymphoma: number analyzed (Participants) | 82
    Lymphoma | 0
    Fluid and electrolyte disorders: number analyzed (Participants) | 82
    Fluid and electrolyte disorders | 7
    Metastatic Cancer: number analyzed (Participants) | 82
    Metastatic Cancer | 0
    Other Neurological Disorders: number analyzed (Participants) | 82
    Other Neurological Disorders | 7
    Obesity: number analyzed (Participants) | 82
    Obesity | 21
    Paralysis: number analyzed (Participants) | 82
    Paralysis | 1
    Peripheral Vascular Disorders: number analyzed (Participants) | 82
    Peripheral Vascular Disorders | 9
    Psychoses: number analyzed (Participants) | 82
    Psychoses | 5
    Pulmonary Circulation disorders: number analyzed (Participants) | 82
    Pulmonary Circulation disorders | 1
    Renal Failure: number analyzed (Participants) | 82
    Renal Failure | 8
    Solid Tumor without Metastasis: number analyzed (Participants) | 82
    Solid Tumor without Metastasis | 7
    Peptic ulcer disease excluding bleeding: number analyzed (Participants) | 82
    Peptic ulcer disease excluding bleeding | 1
    Valvular Disease: number analyzed (Participants) | 82
    Valvular Disease | 9
    Weight Loss: number analyzed (Participants) | 82
    Weight Loss | 1
Immunosuppressive treatments 6 months prior to date of COVID-19 diagnosis [Count of Participants; unit: Participants] — Population: Medical record and claims data were not available for all infused participants to identify a 6 month history of immunosuppressive treatments. The measure provides context for the outcome measures and was not an eligibility criteria.
  Participants
    number analyzed (Participants) | 117
    Received Immunosuppressive Treatment 6 months prior | 1
    Did Not Receive Immunosuppressive Treatment 6 months prior | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of COVID-19 Related Hospitalization at Day 28
Description: Binary outcome; 1 if participants have one or more COVID-19 related hospitalizations during Days 1-28 after at-home infusion, and 0 otherwise
Time Frame: Days 1-28 after at-home infusion of Bamlanivimab
Population: All eligible participants for primary outcome analysis
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Participants testing positive for COVID-19 who received One-time at-home infusion of 700 mg Bamlanivimab
Arm/Group | Treatment
Number analyzed (Participants) | 138
Participants | 6

2. Secondary Outcome: Safety - Documenting Adverse Events After Infusion
Description: Describe the incidence of infusion reactions recorded by the Optum Infusion nurse on the Case Report Form (CRF) during receipt of infusion and during the defined infusion follow-up period. The reporting includes all-cause mortality, COVID-19 related hospitalizations, and all-cause emergency room (ER) visits.
Time Frame: Days 1-28 after at-home infusion of Bamlanivimab
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 138
Participants
  COVID-19 related hospitalization | 6
  All-Cause ER visits | 4

ADVERSE EVENTS:
Time Frame: Days 1-28 after at-home infusion of Bamlanivimab
Description: The reporting includes all-cause mortality, COVID-19 related hospitalizations, and all-cause emergency room (ER) visits. All adverse events were considered serious.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 1/139
Serious Adverse Events (participants affected / at risk) | 10/139
Other Adverse Events (participants affected / at risk) | 0/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=139)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (General disorders) | 1 (1) — participant fainted at start of infusion. Infusion was stopped and participant went to ER. Was discharged without being admitted
Hypokalemia (General disorders) | 1 (1)
Dysarthria (General disorders) | 1 (1) — Participant had shaking, slurring of speech, weakness, and itching and was referred to Emergency Department. Became stable and continued to improve after discharge
Shaking (General disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Shorness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Participant had shortness of breath, increased coughing and febrile. Hospitalized overnight and discharged with improvement
Increased Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT04656691/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT04656691/SAP_003.pdf